CLINICAL TRIAL: NCT01493219
Title: MMP-2, MMP-9 and NGAL as Biomarkers for Glioblastoma (GBM) Biomarkers for the Prognosis of Glioblastoma
Brief Title: Biomarkers for Prognosis of Glioblastoma (GBM)
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0369-11-FB
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Glioblastoma Multiforme; Astrocytoma; Gliosarcoma; Glioma WHO grade IV
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Gliosarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood, Urine, and Tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epilepsy: Blood and urine sample collection, pre and post op
- Glioma: Blood and urine sample collection, pre and post op

SUMMARY:
The purpose of this study is:

1. To learn if (MMP-2, MMP-9 and NGAL) which are substances found in blood and urine associated with tumors, can be used as tumor markers in the management and treatment of glioblastoma.
2. To study the relationship between MMP-2, MMP-9 and NGAL with quality of life and disease symptoms.

DETAILED DESCRIPTION:
Matrix metalloproteinases (MMP) -2 and -9 belong to a multigene family of degradative enzymes implicated in the neoangiogenesis required for tumor growth. In the central nervous system (CNS), MMP-2, MMP-9 and neutrophil gelatinase-associated lipocalin (NGAL) are overexpressed in orthotopic models and also in human brain tumor specimens. Furthermore, serum and urinary levels of these markers have been shown to correlate with the presence and status of brain tumors in all types of primary brain tumors. A major challenge in the treatment of primary brain tumors is the dependence on magnetic resonance imaging (MRI) to differentiate disease progression from treatment-related change. This is particularly challenging in glioblastomas (GBM) where multimodality therapy with radiation and chemotherapy is commonly used and can lead to pseudoprogression and treatment-related tissue necrosis, both of which can masquerade as true tumor progression. Often we are faced with the decision to treat based on imaging findings alone or to recommend that patients have another invasive surgery. We hypothesize that MMP-2, MMP-9 and NGAL will: 1) be detected on tumor tissue by immunohistochemistry and not on non-tumor (epilepsy) brain tissue, 2) parallel the course of disease in the urine and/or serum of patients and 3) remain unchanged in the event of pseudoprogression and treatment related imaging changes. Quality of life, patient symptoms, and cognitive function are vitally important in patients with GBM. Quality of life and selected symptoms will also be assessed and correlated with serum and urine biomarkers. We hope to confirm the utility of MMP-2, MMP-9 and NGAL in the management of GBM.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled for a surgical excision or biopsy as ordered by his/her clinic or inpatient physician for epilepsy OR subjects newly diagnosed with high grade (grade IV) glioma (The performance of this procedure will be under standard of care surgical guidelines.)

   * non-tumor tissue controls from subjects undergoing surgery for epilepsy
   * tumor tissue from subjects undergoing surgery for grade IV glioma
2. Epilepsy subject identified as a control undergoing surgery must willingly provide pre-op and post-op serum and urine samples for research
3. GMB subject must willingly provide blood and urine samples pre-op and post-op as well as blood and urine samples for research and QOL measurements taken at protocol specific time points
4. GBM subject plans to receive clinical care visits which coincide with MRIs and/or with a change in symptoms and any secondary surgical resections and/or biopsies solely at UNMC/TNMC
5. Subjects must willingly give signed informed consent
6. Age 19 years or older (the age of consent in Nebraska)
7. Women must not be pregnant due to teratogenic effects of MRI

Exclusion Criteria:

1. Inability to fulfill the requirements of the protocol
2. No serious disease or condition that, in the opinion of the investigator, would compromise the patient's ability to participate in the study
3. Known to be positive for HIV or infectious hepatitis, type A, B or C or active Hepatitis
4. Subjects newly diagnosed with high grade (grade IV) glioma (GBM) unable to be followed by MRI due to

   * Pacemaker
   * Chronic kidney disease stage 3-5 (Glomerular Filtration Rate <60)
   * Unable to lay flat for 90 minutes
   * Any metallic foreign body not approved for MRI
   * Known hypersensitivity to Gadolinium contrast or other required for MRI

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled for a surgical excision or biopsy as ordered by his/her clinic or inpatient physician for epilepsy OR subjects newly diagnosed with high grade (grade IV) glioma
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-09-20 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
1) To provide preliminary evidence that MMP-2 and MMP-9/NGAL ratio in tissue corresponds with their presence in the urine and blood in patients undergoing surgery for epilepsy (Aim 1a) and in patients with grade IV glioma (Aim 1b) | Up to 3 years
  For each outcome (MMP-2, MMP-9 and MMP-9/NGAL), Pearson's correlation coefficient will be used to examine the association between 1) tissue and urine and 2) tissue and blood. Spearman's correlation will be used in the event that the data are not normally distributed and a suitable transformation is not evident. Due to the anticipated interaction of group with presence of these biomarkers, these analyses will be conducted separately for epilepsy control patients and GBM patients.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole A Shonka, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided